CLINICAL TRIAL: NCT00571636
Title: Efficacy and Safety of Continuous Infusion of Fentanyl for Pain Control in Preterm Newborn on Mechanical Ventilation
Brief Title: Continuous Infusion of Fentanyl in Preterm on MV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Ancora Gina, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEO 01/2005; FARM63TMS3
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Pain; Infant, Premature, Diseases; Respiration; Insufficient or Poor, Newborn
Keywords: Opioids infusion; mechanical ventilation
MeSH Terms: conditions — Pain; Infant, Premature, Diseases; Respiratory Aspiration | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fentanyl (Active Comparator): Patients assigned to this arm will receive continuous infusion of fentanyl + open label boluses of Fentanyl if necessary.
  Interventions: Drug: Fentanyl
- placebo (Placebo Comparator): Patients assigned to this arm will receive continuous infusion of placebo+ open label boluses of Fentanyl if necessary.
  Interventions: Drug: 5% glucose solution

INTERVENTIONS:
Drug: Fentanyl — The experimental drug will be diluted according to each NICU scheme and administered as an attach dose of 1 mcg/kg in 30' followed by continuous i.v. infusion of 1 mcg/kg/h. Infusion of the experimental drug has to begin within 24 hrs from the beginning of MV and has to be continued until the end of MV and not after 7 days of life. If the newborn is still on MV after the 7th day of life he/she will be treated for pain according to local protocols.
  Open label boluses of Fentanyl during the study phase will be administered, in both groups when the EDIN pain score is > 6 and before performing the following invasive procedures:Peripherally inserted central venous catheter positioning;Re-intubation;Lumbar puncture;Pneumothorax or hydrothorax drainage.
  Arms: fentanyl
Drug: 5% glucose solution — ev continuous infusion
  Arms: placebo

SUMMARY:
The objective of this randomized, double-blind trial is to compare the efficacy and safety of 2 therapeutic regimens of fentanyl administration in a population of preterm newborns of GA <= 32 weeks in MV:

* Group A) continuous infusion of Fentanyl + open label boluses of Fentanyl;
* Group B) continuous infusion of placebo + open label boluses of Fentanyl.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the analgesic superiority of Fentanyl given as 'continuous infusion + boluses' versus 'boluses alone' by comparing pain scores obtained by the application of validated algometric scales for chronic pain (EDIN - Echelle Douleur Inconfort Nouveau-Nè) and acute pain (PIPP- Premature Infant Pain Profile).

The secondary objective of the study is to evaluate the safety equivalence of the above 2 therapeutic regimens by recording:

* Rate of mechanically ventilated newborns at one week of age
* Age at which neonates will reach total enteral feeding
* Age (hours) of first meconium passage
* Incidence of intraventricular haemorrhage (IVH), periventricular leucomalacia (PVL) or death within 28 days of life
* Incidence of bladder globe during the first week of life
* Incidence of hypotension during the first week of life

5.2.1 Pain measurement: during the study phase acute pain will be measured once a day during a heel prick by a validated algometric scale for acute pain (PIPP); chronic pain will be measured 3 times a day by a validated algometric scale for chronic pain (EDIN). Inter-rater reliability has been shown acceptable for both scales (26,27). Moreover, in October 2006 the Coordinating Center organized a theoretical and practical course on the correct application of the PIPP and EDIN scales (26,27) for all the participating centers in order to reduce the inter-Center variability in pain measurement.

The EDIN scores will be recorded in a specific CRF (CRF N°1, p. 15). The PIPP scores will be reported in a specific CRF (CRF N° 1, pp. 8-14).

5.2.2 Painful procedures: the following painful procedures, as well as the action taken to reduce pain, will be recorded in the same CRF (CRF N° 1, pp. 8-14):

* heel pricks
* endotracheal aspirations
* venous blood samplings
* pneumothorax drainage
* peripherally inserted central catheter positioning
* others (specify) 5.2.3 Fentanyl open label boluses administration: all the boluses of open label fentanyl administered according to the criteria reported in paragraph 6.1.1 have to be recorded in a special CRF (CRF N° 1, p. 7).

5.2.4 Instrumental examinations: a heart ultrasound has to be obtained in all newborns in the first week of life in order to diagnose patent ductus arteriosus. Brain ultrasound has to be repeated at 4, 7 days of age and then twice a month or when clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* inborn neonates
* preterm neonates ≤ 32+ 6 days weeks gestation
* < 72 hours of life
* newborns on MV
* within 24 hours from the beginning of MV administered through an endotracheal tube
* parental written informed consent for participation in the study must be obtained

Exclusion Criteria:

* Evidence of severe birth asphyxia, that is an APGAR score below 4 at 5 minutes of age and/or umbilical arterial pH < 7.0
* Known genetic or chromosomal disorders
* Severe IVH (> grade II according to Volpe classification (30))
* Need for post-operative analgesic therapy in the first week of life
* Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable for this study will be the pain scores obtained during the study period. Procedural pain will be measured once a day by the PIPP scale. Chronic pain will be evaluated through the application of the EDIN scale 3 times a day. | 7 days

SECONDARY OUTCOMES:
Rate of MVd newborns at one week of age;Age at which neonates will reach total enteral feeding;Age of first meconium passage;Incidence of IVH, PVL or death within 28 days of life;Incidence of bladder globe and hypotension during the first week of life | until discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Gina Ancora, Doctor, Principal Investigator — St'Orsola-Malpighi General Hospital
Locations (1):
- St'Orsola-Malpighi General Hospital, Bologna, BO, Italy

REFERENCES:
- [Derived] Ancora G, Lago P, Garetti E, Pirelli A, Merazzi D, Mastrocola M, Pierantoni L, Faldella G. Efficacy and safety of continuous infusion of fentanyl for pain control in preterm newborns on mechanical ventilation. J Pediatr. 2013 Sep;163(3):645-51.e1. doi: 10.1016/j.jpeds.2013.02.039. Epub 2013 Apr 10. PMID 23582138